CLINICAL TRIAL: NCT02557009
Title: Changes in Hemodynamic Values With Posture
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Kane High, Associate Professor, Milton S. Hershey Medical Center
Other Study IDs: 044000EP
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Blood Pressure
Keywords: Hemodynamics; Central Venous Pressure; Pulmonary Artery Pressure; Cardiac Output

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is designed as a prospective observational study. Each participant will have their BP, CVP, PAP, and CO measured by their clinical nurse using indwelling catheters placed for routine patient monitoring. Measurements will be recorded on an hourly basis during the day and for as many days as possible if the required measurements are being made for clinical care.

Sixty patients between 18 and 85 years of age will be recruited in HVICU by means of convenience sampling. Data will be analyzed using a test of equivalence on the initial measurements (test of equivalence between two means) and then over time (repeated measurements) with a linear mixed-effects model.

DETAILED DESCRIPTION:
Invasive monitoring is a common method used in intensive care units to measure cardiovascular status. These parameters include central venous pressure (CVP), pulmonary artery pressure (PAP) cardiac output (CO) and arterial blood pressure (BP). There is a general understanding that these parameters vary with the position of the patient with the expectation that, as the patient goes from supine to sitting, these parameters decrease to some extent due to decreased venous return to the heart. Furthermore, the extent to which a patient might be reclining in bed can vary greatly from just having the head slightly raised to being totally upright. Different policies exist with respect to patient position when these measurements are made. The policies vary from no specified position to placing them completely flat for making the measurement and then returning them to a more upright position, usually 30 or 45 degrees. Decisions are based upon the supine measurements despite no clear correlation to the patient's usual position. This study will investigate the correlation between position and these parameters.

Patients in the HVICU will be approached by a member of the research team and asked for their verbal approval to record measurements made by their nurse. After receiving verbal consent to record the measurements, a member of the study team will record BP. CVP, PAP and CO as measured by the patient's nurse. These measurements will be recorded with the patient lying on the bed with the back of the bed raised to 30o and with the patient supine when the back of the bed is at 0o. The transducers will be leveled with the anterior axillary by zeroing of the transducer. After each position change, the team member will ask the nurse to wait 5 minutes to allow stabilization of these parameters before measuring and recording the parameters at that position. These parameters will be recorded on an hourly basis using the day for as many days as the required measurements are being made for clinical care. Other patient information recorded will be date, ejection fraction, BMI, height, weight, age, and PEEP, if the patient is intubated.

Sixty patients between 18 and 85 years of age will be recruited in HVICU by means of convenience sampling. The sample size was calculated based on the initial measurement of CVP where our preliminary data shows a mean difference 1.28±2.93 mmHg, and assuming that values with a difference < 3 are equivalent, with an α = 0.05 and a power of 90. The calculation was done at the following website: http://www.sealedenvelope.com/power/continuous-equivalence. Data will be analyzed using a test of equivalence on the initial measurements (test of equivalence between two means) and then over time (repeated measurements) with a linear mixed-effects model.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18 to 85 years of age) in the HVICU
2. Have indwelling CVP or PA catheter.

Exclusion Criteria:

1. Patients who have just undergone mitral valve surgery
2. Patients that have PEEP > 10cmH2O

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Hershey Medical Center having CABG and aortic valve surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
central venous pressure supine and with head of bed at 30 degrees | 48 hours post-operatively

SECONDARY OUTCOMES:
cardiac output supine | 48 hours post-operatively
cardiac output with head of bed at 30 degrees | 48 hours post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Kane High, MD, Principal Investigator — MS Hershey Medical Center
Locations (1):
- Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania, United States